CLINICAL TRIAL: NCT06193213
Title: Incidence of Postoperative Residual Curarization, a Prospective Observational Study
Brief Title: Incidence of Postoperative Residual Curarization
Acronym: PORC
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 5991
Record Dates: First submitted 2023-12-11; First posted 2024-01-05 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2023-12

CONDITIONS: Neuromuscular Blockade, Residual
MeSH Terms: conditions — Delayed Emergence from Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: measurement of train of four ratio (TOFR) to assess residual neuromuscolar block — Upon arrival of the spontaneously breathing patient in the Post-Anesthesia Care Unit, a researcher will evaluate the TOFR to detect any residual neuromuscular block using the acceleromyographic method at the level of thumb adductor.2 TOFR measurements will be performed 30 seconds apart. If the difference between the two measurements will be ≤ 0.1, the average value will be considered for the purposes of the analysis. In case of a difference > 0.1, a third measurement will be taken and the average of the two closest results will be considered. If a residual block is detected sugammadex will be administered (2 mg/kg in the case of at least 2 contraction responses to TOF stimulation or 4 mg/kg in the case of no contraction response) to restore normal neuromuscular function , assessed by subsequent TOFR measurement.

SUMMARY:
An incomplete postoperative recovery of neuromuscular function (postoperative residual curarization - PORC) represents a common problem in post-anesthesia care units (PACU), potentially exposing the patient to adverse respiratory events.

Quantitative and objective evaluation of neuromuscular function using the train acceleromyographic method -of-four ratio (TOFR) at the level of the adductor muscle of the thumb represents the best way to minimize this risk after administration of non-depolarizing neuromuscular agents.

Study endpoints Primary endpoint

* incidence of postoperative residual curarization Secondary endopoints
* number of possible respiratory adverse events during the stay in the PACU and during the hospital stay
* estimation of a logistic regression model to define the risk factors associated with residual curarization

DETAILED DESCRIPTION:
Neuromuscular blocking agents are commonly used in clinical anesthetic practice to facilitate tracheal intubation and allow muscle relaxation during surgical interventions.

Anesthesiologist's subjective qualitative assessment of the patient's recovery of muscle strength before extubation is not predictive of adequate neuromuscular recovery even if many surveys conducted at an international level [1,2,3] demonstrate how this modality of evaluation is often used above all due to the not always widespread availability of tools for quantitative monitoring of neuromuscular blockade3.

An incomplete recovery of neuromuscular function at the end of surgery (Postoperative residual curarization - PORC) exposes the patient to potential adverse respiratory events and a Consensus Statement [4] of experts in 2018 suggested a quantitative and objective evaluation of neuromuscular function using the train acceleromyographic method -of-four ratio (TOFR) at the level of the adductor muscle of the thumb represents the best way to minimize this risk after administration of non-depolarizing neuromuscular agents.

In case of TOFR ≤ 0.9, reversal of the neuromuscular block is normally performed with drugs belonging to the class of acetylcholinesterase inhibitors (e.g. neostigmine 0.03-0.05 mg/kg, associated with an antimuscarinic agent such as atropine to counteract the cholinergic effects) or by sugammadex (2 or 4 mg/Kg), a selective antagonist of rocuronium and vecuronium which acts by encapsulating the neuromuscular blocking molecule making it ineffective.

Recurrence of neuromuscular blockade may, however, occur primarily due to mechanisms of redistribution of the muscle relaxant or if insufficient doses of the reversal drug are administered.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged ≥ 18 years, American Society of Anesthesiologists (ASA) physical status I-III, who have expressed written consent to participate in the study and who will undergo surgery under general anesthesia with the use of non-depolarizing neuromuscular blocking agents at intermediate duration of action, to facilitate tracheal intubation and/or for maintaining a condition of myoresolution during surgery.

Exclusion Criteria:

* Patients undergoing emergency surgery, who do not require the administration of non-depolarizing neuromuscular blockers, patients with neuromuscular pathologies, or who require postoperative monitoring in the Intensive Care Unit.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing surgery under general anesthesia with the use of non-depolarizing neuromuscular blocking agents at intermediate duration of action, to facilitate tracheal intubation and/or for maintaining a condition of myoresolution during surgery
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
postoperative residual neuromuscular block | within 5 minutes from admission in the postoperative care unit
  evaluation of the incidence of postoperative residual neuromuscular block upon arrival in the post-anesthesia care unit (PACU), defined as a TOFR≤0.9, by acceleromyographic method in interventions in which non-depolarizing neuromuscular blockers with intermediate duration of action were administered at the time of tracheal intubation and/or for maintaining a condition of myoresolution during surgery.

SECONDARY OUTCOMES:
number of respiratory adverse events | within 7 days
  Number of any adverse respiratory events that occurred during the stay in the PACU and during the hospital stay. Respiratory adverse events will be defines as episodes of desaturation (SpO2<92%) requiring oxygen supplementation or the finding of atelectasis, pneumonia or pleural effusion of non-cardiac origin found on thoracic imaging tests possibly performed during the hospital stay;
evaluation of possible risk factors for residual curarization | 4 months
  Estimation of a logistic regression model to define risk factors for residual curarization Will be considered as possible risk factors those reported in the literature : the patient's age, the duration of anesthesia, the type of anesthesia administered (inhalation or totally intravenous), the number of administrations and the total dose of neuromuscular blocker, reversal or not of the neuromuscular blockade, the antagonist drug and the type of neuromuscular blocker used during surgery [7].

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Piersanti, MD, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Piersanti A, Garra R, Sbaraglia F, Del Vicario M, Lamacchia R, Rossi M. Neuromuscular monitoring and incidence of postoperative residual neuromuscular blockade: a prospective observational study. J Anesth Analg Crit Care. 2025 Jan 28;5(1):5. doi: 10.1186/s44158-025-00226-1. PMID 39875976

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-23): https://cdn.clinicaltrials.gov/large-docs/13/NCT06193213/Prot_SAP_000.pdf